CLINICAL TRIAL: NCT00980694
Title: Bioavailability of Ubiquinol in Huntington Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Kaneka Corporation (Industry)
Responsible Party: Principal Investigator, Karl Kieburtz, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UQ01
Record Dates: First submitted 2009-09-17; First posted 2009-09-21 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Huntington Disease
Keywords: ubiquinol; coenzyme Q10; Huntington disease
MeSH Terms: conditions — Huntington Disease | interventions — ubiquinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ubiquinol (Experimental): up to 600 mg per day, oral capsules for 8 weeks
  Interventions: Dietary Supplement: ubiquinol

INTERVENTIONS:
Dietary Supplement: ubiquinol — up to 600 mg per day, oral capsules for 8 weeks

SUMMARY:
The death of brain cells in Huntington Disease (HD) is thought to be associated with a lack of normal cell energy and harmful brain substances called free radicals. Coenzyme Q10 (CoQ) is a marketed nutritional supplement that may prove useful in HD because it increases cell energy and combats free radicals.

Most studies of CoQ have looked at only one formulation of CoQ ("ubiquinone") in HD. The purpose of the study is to find out if people that switch from the common formulation of CoQ ("ubiquinone") to a different formulation ("ubiquinol") have higher levels of CoQ in their blood after taking the same dose. The investigators also want to find out if this different formulation is tolerable for individuals with HD.

ELIGIBILITY:
Inclusion Criteria:

* Have manifest Huntington disease
* Be 18 years of age or older
* Be taking an oxidized formulation of CoQ for at least 30 days prior to the baseline visit
* Be on a steady dose of all concomitant medications for at least 30 days prior to the baseline visit

Exclusion Criteria:

* Have a history of intolerability of sensitivity to CoQ
* Have an unstable medical or psychiatric illness
* Be pregnant or breastfeeding; women of childbearing age must use reliable contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
serum coenzyme Q10 levels | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karl Kieburtz, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States